CLINICAL TRIAL: NCT02388516
Title: Maternal Vitamin D for Acute Respiratory Infections in Infancy (MDARI): a Nested Sub-study in a Randomized Controlled Trial of Vitamin D Supplementation During Pregnancy and Lactation in Dhaka, Bangladesh
Brief Title: Maternal Vitamin D for Acute Respiratory Infections in Infancy
Acronym: MDARI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, Daniel Roth, Clinician-Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1000039072-ARI
Record Dates: First submitted 2015-03-09; First posted 2015-03-17 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Upper Respiratory Tract Infections; Lower Respiratory Tract Infections
Keywords: Bangladesh; Vitamin D; Acute Respiratory Infections; Infancy; Pregnancy
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group A (Placebo Comparator): Prenatal Period 0 IU; Postpartum Period 0 IU (placebo) Overall: The Prenatal Period will start at enrolment (17-24 weeks gestation) and last until delivery. The Postpartum Period will last from delivery until 6 months postpartum.
  Interventions: Dietary Supplement: Placebo
- Group B (Experimental): Prenatal Period 4,200 IU/week of vitamin D3; Postpartum Period 0 IU/week (placebo)
  Interventions: Dietary Supplement: Vitamin D3
- Group C (Experimental): Prenatal Period 16,800 IU/week of vitamin D3; Postpartum Period 0 IU/week (placebo)
  Interventions: Dietary Supplement: Vitamin D3
- Group D (Experimental): Prenatal Period 28,000 IU/week of vitamin D3; Postpartum Period 0 IU/week (placebo)
  Interventions: Dietary Supplement: Vitamin D3
- Group E (Experimental): Prenatal Period 28,000 IU/week of vitamin D3; Postpartum Period 28,000 IU/week
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3
  Other Names: Cholecalciferol
  Arms: Group B; Group C; Group D; Group E
Dietary Supplement: Placebo
  Arms: Group A

SUMMARY:
There is a growing body of data suggesting that vitamin D modulates the host's immune response to acute respiratory infection (ARI). The primary aim of this study is to determine whether maternal vitamin D3 supplementation versus placebo decreases the incidence rate of microbiologically confirmed viral-associated ARI among infants in Dhaka, Bangladesh. Secondary outcomes include: A) incidence of ARI associated with specific major pathogens, B) incidence of clinical ARI (without the need for positive microbiology), and C) quantitative density of pneumococcal carriage. Infants will be followed from birth until 6 months of life. Among infants who meet at least one of the specific case definitions for ARI (see 'Detailed Description' section), nasal swab specimens will be collected. Respiratory samples will be analyzed by real-time polymerase chain reaction (qPCR) to identify a 7-virus panel (influenza A and B, respiratory syncytial virus, human metapneumovirus, adenovirus, and parainfluenza types 1, 2, and 3) plus quantitative density of S. pneumonia.

DETAILED DESCRIPTION:
In this study, an acute respiratory infection (URTI and/or LRTI) has been clinically defined as:

A) Upper respiratory tract infection (URTI)

A new-onset illness consisting of at least two of the following clinical criteria at any time during a surveillance week:

* Caregiver-reported cough;
* Caregiver-reported rhinorrhea;
* Caregiver-reported nasal congestion; and,
* Measured axillary temperature greater than or equal to 37.5°C.

B) Lower respiratory tract infection (LRTI)

1. New onset clinically-diagnosed LRTI:

   * Caregiver-reported cough AND/OR difficulty breathing during a surveillance week; AND,
   * Observed lower chest wall indrawing AND/OR elevated respiratory rate (60 breaths per minute or greater for infant up to 59 days of age, or 50 breaths per minute or greater for infant 60 days of age or older)
2. Hospitalized LRTI

   * Hospitalization with physician diagnosis of pneumonia or bronchiolitis

ELIGIBILITY:
Inclusion Criteria:

* Infants born to women enrolled in the MDIG trial (NCT01924013).
* Maternal inclusion criteria (at time of enrolment) will be:
* At least 18 years of age
* 17 to 24 completed weeks of gestation
* Intends to permanently reside in the trial catchment area for at least 18 months
* Family plans to reside in catchment area for the first 6 months postnatal
* Provides written informed consent for participation

Exclusion Criteria:

* Mother withdrawn from MDIG trial prior to delivery
* Failure to provide consent for participation in sub-study

Ages: 1 Day to 26 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1214 (Actual)
Dates: Start 2014-12; Primary Completion 2016-08-21 (Actual); Study Completion 2016-08-21 (Actual)

PRIMARY OUTCOMES:
Microbiologically confirmed viral acute respiratory infection (URTI and/or LRTI) | 0 to 6 months

SECONDARY OUTCOMES:
ARI with microbiologically confirmed influenza A or B | 0 to 6 months
ARI with microbiologically confirmed RSV | 0 to 6 months
Clinical URTI and/or LRTI (i.e., no microbiological confirmation) | 0 to 6 months
Clinical URTI (i.e., no microbiological confirmation) | 0 to 6 months
Clinical LRTI (i.e., no microbiological confirmation) | 0 to 6 months
Quantitative S. pneumoniae nasal carriage density | 0 to 6 months
Pneumonia (non-severe) and severe pneumonia or very severe disease | 2 to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shaun K Morris, MD, MPH, Principal Investigator — The Hospital for Sick Children; Daniel Roth, MD, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangldesh, Dhaka, Bangladesh

REFERENCES:
- [Derived] Taghivand M, Pell LG, Rahman MZ, Mahmud AA, Ohuma EO, Pullangyeum EM, Ahmed T, Hamer DH, Zlotkin SH, Gubbay JB, Morris SK, Roth DE. Effect of maternal vitamin D supplementation on nasal pneumococcal acquisition, carriage dynamics and carriage density in infants in Dhaka, Bangladesh. BMC Infect Dis. 2022 Jan 13;22(1):52. doi: 10.1186/s12879-022-07032-y. PMID 35026987
- [Derived] Morris SK, Pell LG, Rahman MZ, Dimitris MC, Mahmud A, Islam MM, Ahmed T, Pullenayegum E, Kashem T, Shanta SS, Gubbay J, Papp E, Science M, Zlotkin S, Roth DE. Maternal vitamin D supplementation during pregnancy and lactation to prevent acute respiratory infections in infancy in Dhaka, Bangladesh (MDARI trial): protocol for a prospective cohort study nested within a randomized controlled trial. BMC Pregnancy Childbirth. 2016 Oct 13;16(1):309. doi: 10.1186/s12884-016-1103-9. PMID 27737646